CLINICAL TRIAL: NCT03622775
Title: Daratumumab-Based Maintenance in Patients With Relapsed Multiple Myeloma After Salvage Autologous Stem Cell Transplantation
Brief Title: Daratumumab in Treating Participants With Relapsed Multiple Myeloma After Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0681; NCI-2018-01432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0681 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-16; First posted 2018-08-09 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab) (Experimental): Beginning 60-120 days after transplant, participants receive daratumumab IV over 4-8 hours on days 1, 8, 15 and 22 of courses 1 and 2 and days 1 and 15 of courses 3-6, then on day 1 of subsequent courses. Courses repeat every 28 days for 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414

SUMMARY:
This phase II trial studies whether daratumumab and hyaluronidase-fihj and pomalidomide work in treating patients with multiple myeloma that has come back (relapsed) after stem cell transplant. Daratumumab and hyaluronidase-fihj is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as pomalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving daratumumab and hyaluronidase-fihj with pomalidomide may help control the disease in patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the complete remission rate (CRR) by the International Myeloma Working Group (IMWG) criteria within 9 months post salvage auto-transplant with subcutaneous daratumumab and hyaluronidase-fihj plus pomalidomide maintenance therapy starting approximately 3 months post salvage auto-transplant in patients with relapsed myeloma.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS).

EXPLORATORY OBJECTIVES:

I. To discover the impact of daratumumab and hyaluronidase-fihj plus pomalidomide on graft function and immune reconstitution.

OUTLINE:

Beginning 60-180 days after transplant, patients daratumumab and hyaluronidase-fihj subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6, and then on day 1 of subsequent cycles. Patients also receive pomalidomide orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have had relapsed disease prior to transplant, or undergone previous autologous stem cell transplant (ASCT), followed by relapse and at least a partial response to salvage therapy
* Eligible patients will be enrolled in the protocol no less than 60 days and must be initiated no longer than 180 (+/- 14) days post autologous stem cell transplantation (ASCT)
* Male or female patients 18 years or older.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Patients' clinical laboratory values and toxicity must be as specified below within 14 days before the first dose of the study drug:

  * Platelet count >= 50,000/mm^3
  * Absolute neutrophil count >= 1000/ mm^3 (no growth factors within 5 days)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3 x upper limit of normal (ULN)
  * Creatinine <= 2.5 mg/dL
  * Recovered (i.e., =< grade 2 toxicity) from the reversible effects of autologous stem cell transplant
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care must be obtained, with the understanding that consent may be withdrawn by the subject at any time without any prejudice to future medical care
* Left ventricular ejection fraction >/=40% at the patient's last recorded echocardiogram (this could refer to pretransplant ECHO. ECHO may be repeated if the PI considers a repeat ECHO). No uncontrolled arrythmias.

Exclusion Criteria:

* Major surgery within 14 days before the first dose of study drug
* Radiotherapy within 14 days before enrollment
* Non-secretory disease, plasma cell leukemia, or previous allogeneic transplant
* Known active central nervous system involvement
* Inability or unwillingness to comply with the drug administration requirements
* Female subject is pregnant or lactating
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Patients with a known history of asthma or chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal.
* Patients with moderate or severe persistent asthma within the past 2 years and currently uncontrolled asthma of any classification.
* Infection requiring IV systemic antibiotic therapy within 7 days before cycle day 1 (C1D1) of therapy
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations
* Failure to have fully recovered (i.e., <= grade 2 toxicity) from the effects of prior chemotherapy regardless of the interval since last treatment
* Patient is refractory or resistant to daratumumab and pomalidomide
* Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* If patient was unable to tolerate daratumumab or pomalidomide in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H Qazilbash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.: Beginning 60 days to 180 (+/- 14) days post ASCT, patients with relapsed multiple myeloma prior to transplant, or undergone previous ASCT, followed by relapse and at least a partial response to salvage therapy will receive maintenance therapy with daratumumab/hyaluronidase-fihj and pomalidomide.
  Daratumumab 1800 mg/hyaluronidase-fihj 30,000 units will be given SC weekly for weeks 1-8, followed by every 2 weeks for weeks 9-24, and then every month for weeks 25 until progression.
  Pomalidomide will be given at 2 mg PO daily from day 1-21 in the 28-day cycle for up to 4 weeks.
Period: Overall Study
Arm/Group | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission
Description: Number of participants that achieved Complete remission (CR) 9 months post auto transplant.
  Complete remission (CR) (all of the following):
  1. Negative immunofixation in serum and urine.
  2. < 5% plasma cells in the bone marrow.
  3. Disappearance of any soft tissue plasmacytomas.
Time Frame: Within 9 months post salvage auto transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.
Number analyzed (Participants) | 13
Participants | 11

2. Secondary Outcome: Number of Participants That Relapsed With Progression-free Survival (PFS)
Description: Progression-free survival is defined as the interval from the date of initiation of maintenance therapy after salvage ASCT to the earlier of the first documentation of objective disease progression or death from any cause.
Time Frame: From the date of initiation of maintenance therapy assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.
Number analyzed (Participants) | 13
Participants
  PFS at 20 months | 11
  PFS at 36 months | 8
  PFS at 60 months | 7

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients.
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients. (N=13)
ALT increased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1)
Low granulocyte (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Therapy With Daratumumab/Hyaluronidase-fihj/Pomalidomide Post ASCT in MM Patients. (N=13)
(Investigations) | 1 (1)
(Metabolism and nutrition disorders) | 1 (1)
(Musculoskeletal and connective tissue disorders) | 1 (2)
(Respiratory, thoracic and mediastinal disorders) | 1 (1)
(Musculoskeletal and connective tissue disorders) | 1 (1)
(Respiratory, thoracic and mediastinal disorders) | 1 (2)
ALK increased (Investigations) | 1 (2)
ALT increased (Investigations) | 4 (4)
Anemia (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
AST increased (Investigations) | 2 (2)
Bacterial (Infections and infestations) | 4 (5)
Bacterial (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Edema (General disorders) | 4 (5)
Fatigue (General disorders) | 6 (11)
Hypogammaglobulinemia (Immune system disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5)
LDH increased (Investigations) | 2 (2)
Low granulocyte (Blood and lymphatic system disorders) | 5 (11)
Low platelet (Investigations) | 5 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 7 (49)
(Renal and urinary disorders) | 1 (1)
(Skin and subcutaneous tissue disorders) | 1 (2)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
T bilirubin increased (Investigations) | 1 (1)
Viral (Infections and infestations) | 7 (20)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wbc decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT03622775/Prot_SAP_001.pdf
  • Informed Consent Form (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT03622775/ICF_000.pdf